CLINICAL TRIAL: NCT00627887
Title: Randomised Controlled Trial of Electroconvulsive Therapy (ECT) With Pharmacotherapy or Pharmacotherapy Alone in Relapse Prevention of Depression
Brief Title: Randomised Controlled Trial of Electroconvulsive Therapy (ECT) in Relapse Prevention of Depression
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Örebro County Council (Other Government)
Collaborators: Uppsala-Örebro Regional Research Council (Other)
Responsible Party: Principal Investigator, prof Ingemar Engström, Professor, Örebro County Council
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ISRCTN40355220; ISRCTN40355220
Record Dates: First submitted 2008-01-04; First posted 2008-03-04 (Estimated); Last update posted 2012-06-22 (Estimated); Status verified 2012-06

CONDITIONS: Depressive Disorder, Major
Keywords: Depressive Disorder, Major; Electroconvulsive Therapy; Lithium Carbonate; venlafaxine
MeSH Terms: conditions — Depressive Disorder, Major | interventions — Electroconvulsive Therapy; Venlafaxine Hydrochloride; Lithium; Lithium Carbonate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- ECT+pharmacotherapy (Experimental): Unilateral brief pulse ECT weekly for 6 weeks thereafter every 2 weeks; Venlafaxine target dose 300mg/day; Lithium target dose 0,5-0,8 mmol/L.
  Interventions: Procedure: Electroconvulsive therapy; Drug: venlafaxine; Drug: Lithium
- pharmacotherapy (Active Comparator): Venlafaxine target dose 300mg/day; Lithium 0,5-0,8 mmol/L.
  Interventions: Drug: venlafaxine; Drug: Lithium

INTERVENTIONS:
Procedure: Electroconvulsive therapy — unilateral briefpulse ECT weekly for the first 6 weeks thereafter every 2 weeks for a total of one year
  Other Names: ECT
  Arms: ECT+pharmacotherapy
Drug: venlafaxine — extended release target dose of 300mg/day duration of one year
  Other Names: Efexor; Effexor
Drug: Lithium — serum concentration 0,5-0,8 mmol/L, one year duration
  Other Names: Lithionit; Lithobid; Eskalith

SUMMARY:
The purpose of the study is to determine if continuation electroconvulsive therapy (ECT) is safe and effective in relapse prevention of depression.

DETAILED DESCRIPTION:
Randomized multicenter clinical trial with two parallel groups. Patients with major depression (unipolar or bipolar), who have remitted with electroconvulsive therapy (ECT) are eligible. All patients receive pharmacotherapy (venlafaxine target dose 300mg/day, and lithium target dose 0,5-0,8 mmol/L). The intervention is continuation unilateral ECT weekly for the first 6 weeks thereafter every 2 weeks for one year. Depressive relapse is the primary outcome measure.

ELIGIBILITY:
Inclusion Criteria:

1. MINI-PLUS verified major depressive episode (unipolar or bipolar).
2. ECT within the last 3 weeks.
3. Either Remission defined as MADRS < 10 or
4. Response defined as MADRS < 15 combined with patient assessed CGI-I of at least much improved

Exclusion Criteria:

1. Schizophrenia or Schizoaffective disorder
2. Addiction or Dependence
3. Kidney disease that contraindicates lithium treatment
4. Vascular or heart disease that contraindicates venlafaxine treatment
5. Uncontrolled Epilepsia
6. Age less that 18
7. Pregnancy or Lactation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2008-01; Primary Completion 2012-05 (Actual); Study Completion 2012-05 (Actual)

PRIMARY OUTCOMES:
MADRS >20, psychiatric hospitalization or suicide | 1 year, all patients assessed if MADRS-S > 20 and at 2,6 and 12 months

SECONDARY OUTCOMES:
Mini Mental State Examination | 2,6 and 12 months
ADAS-cog | 2,6 and 12 months
Autobiographical Memory Inventory -Short Form (AMI-SF) | 2,6 and 12 months patients treated in Örebro
Clinical Global Impression-Severity | 2,6 and 12 months
Udvalg for Kliniske Undersogelser (UKU) | 2, 6 and 12 months
MADRS-S Montgomery Asberg Depression Rating scale- self assessment | weekly for 6 weeks thereafter every 2 weeks for a total of one year

CONTACTS AND LOCATIONS:
Overall Officials: Ingemar Engstrom, MD, PhD, Principal Investigator — County Council of Orebro, University of Orebro, Sweden; Axel Nordenskjold, MD, Study Director — County Council of Orebro,; Lars von Knorring, PhD, MD, Study Director — County Council of Uppsala, University of Uppsala Sweden
Locations (4):
- Sweden (4):
  - Psychiatric Clinic, Säter, Dalarna County
  - Löwenströmska sjukhuset, Stockholm, Stockholm County
  - Psychiatric Clinic, Uppsala, Uppsala County
  - Psychiatric clinic, Örebro, Örebro County

REFERENCES:
- [Background] Kellner CH, Knapp RG, Petrides G, Rummans TA, Husain MM, Rasmussen K, Mueller M, Bernstein HJ, O'Connor K, Smith G, Biggs M, Bailine SH, Malur C, Yim E, McClintock S, Sampson S, Fink M. Continuation electroconvulsive therapy vs pharmacotherapy for relapse prevention in major depression: a multisite study from the Consortium for Research in Electroconvulsive Therapy (CORE). Arch Gen Psychiatry. 2006 Dec;63(12):1337-44. doi: 10.1001/archpsyc.63.12.1337. PMID 17146008
- [Background] Sackeim HA, Haskett RF, Mulsant BH, Thase ME, Mann JJ, Pettinati HM, Greenberg RM, Crowe RR, Cooper TB, Prudic J. Continuation pharmacotherapy in the prevention of relapse following electroconvulsive therapy: a randomized controlled trial. JAMA. 2001 Mar 14;285(10):1299-307. doi: 10.1001/jama.285.10.1299. PMID 11255384
- [Derived] Brus O, Cao Y, Carlborg A, Engstrom I, von Knorring L, Nordenskjold A. Long-Term Effect of Maintenance Electroconvulsive Therapy in Patients With Depression-Data From a Small Randomized Controlled Trial. J ECT. 2024 Sep 1;40(3):169-172. doi: 10.1097/YCT.0000000000000983. Epub 2023 Dec 28. PMID 38232249
- [Derived] Nordenskjold A, von Knorring L, Ljung T, Carlborg A, Brus O, Engstrom I. Continuation electroconvulsive therapy with pharmacotherapy versus pharmacotherapy alone for prevention of relapse of depression: a randomized controlled trial. J ECT. 2013 Jun;29(2):86-92. doi: 10.1097/YCT.0b013e318276591f. PMID 23303421